CLINICAL TRIAL: NCT01626508
Title: Directed Donation of Untreated Milk or Milk Processed by the Breast-milk : Prospective Evaluation in Older Premature
Brief Title: Prospective Evaluation in Older Premature, Untreated Breast Milk and Milk Processed by the Breast-milk Bank
Acronym: ADiLL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Collaborators: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: IACOBELLI PHRC IR 2011
Record Dates: First submitted 2012-06-18; First posted 2012-06-22 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Infant, Premature, Diseases; Fatty Acid Deficiency
Keywords: breast milk; breast-milk bank; plasma profile; essential fatty acids
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample milk
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- breast-milk bank: breast milk collected and processed by the breast-milk bank before being used
- breast milk: breast milk used without any treatment, directly by children

SUMMARY:
The purpose of this study is to evaluate the impact of the enteral nutrition type (untreated breast milk, or breast milk processed by the breast-milk bank) on the longitudinal evolution of the total content and plasma profile of essential fatty acids (EFA) in a population of premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Parent's written informed consent
* Gestational age less than 33 weeks of amenorrhea
* Hospitalisation in an NICU at the time of inclusion
* Intended enteral nutrition with breast milk

Exclusion Criteria:

* Persons not covered by the French social security system
* Major congenital malformation
* Participation in other biomedical study protocols
* Babies that are likely to be transferred to another hospital during the study period

Ages: 1 Minute to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: for both groups, the gestational age at birth must be less than 33 weeks gestation and at the time of inclusion the child must be hospitalized in neonatal resuscitation
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Measurement of the effects of the milk-treatment process at the milk bank on the composition of the milk in terms of FA | 3 weeks after the establishment of enteral nutrition
  * Level of total FA and composition of FA on samples of untreated breast milk immediately after the milk has been expressed
  * Level of total FA and composition of FA on samples of breast milk provided by the milk bank just before being given to the infant

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire, Dijon, Bourgogne-Franche-Comté
  - Centre Hospitalier Regional, Saint-Pierre, LA Reunion